CLINICAL TRIAL: NCT04429737
Title: Department of Traditional Chinese Medicine, Keelung Chang Gung Memorial Hospital
Brief Title: The Effects of Freshwater Clam Extract on Blood Sugar, and Lipid Profile in Prediabetes Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Zhao Hong Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Chang Gung IRB 201601965A3
Record Dates: First submitted 2020-05-05; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-05

CONDITIONS: Prediabetes; Metabolic Diseases; Glucose Metabolism Disorders; Dietary Supplement; Nutrition
Keywords: Prediabetes; Glucose Metabolism Disorders; Metabolic Diseases; Clam protein capsules; Clam peptide; Clam amino capsules; clam extract
MeSH Terms: conditions — Prediabetic State; Metabolic Diseases; Glucose Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The prediabetes patients in this arm will receive Clam protein capsules or Clam peptide plus Chlorella capsules with a dose for 2g/d (500mg/capsule, 2 capsules/time, 2 times/day at day and night ) for 6 months.
  Interventions: Dietary Supplement: clam protein capsules; Dietary Supplement: Clam peptide plus Chlorella capsules
- placebo (Placebo Comparator): The prediabetes patients in this arm will receive placebo with similar appearance of Clam protein capsules or Clam peptide plus Chlorella capsules.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: clam protein capsules — The prediabetes patients in this arm will receive Clam protein capsules with a dose for 2g/d (500mg/capsule, 2 capsules/time, 2 times/day at day and night ) for 6 months ( Blood draw every 3 months) . After taking tested substance 6 months, the prediabetes patients will be continuous tracked for 3 years and be blood drawed every 6 months.
  Arms: Experimental
Dietary Supplement: Clam peptide plus Chlorella capsules — The prediabetes patients in this arm will receive Clam peptide plus Chlorella capsules with a dose for 2g/d (500mg/capsule, 2 capsules/time, 2 times/day at day and night ) for 6 months ( Blood draw every 3 months) . After taking tested substance 6 months, the prediabetes patients will be continuous tracked for 3 years and be blood drawed every 6 months.
  Arms: Experimental
Dietary Supplement: Placebo — The prediabetes patients in this arm will receive Placebo with a dose for 2g/d (500mg/capsule, 2 capsules/time, 2 times/day at day and night ) for 6 months ( Blood draw every 3 months) . After taking tested substance 6 months, the prediabetes patients will be continuous tracked for 3 years and be blood drawed every 6 months.
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether the freshwater clam extract and its combination is effective on the improvement of glucose and lipid metabolism, also evaluate its ability to postpone prediabetes patients to become diabetes.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of freshwater clam extract and its combination is effective on the improvement of glucose and lipid metabolism, as well as evaluate its ability to postpone prediabetes patients to become diabetes., 3 month and 6 month data will be collected and put into analysis to provide some suggestions on the Clam protein capsules and Clam peptide plus Chlorella capsules use in the clinical practice for prediabetes patients.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to cooperate in the trial and sign the written informed consent
2. Age 25-70 years
3. Glucose AC between 100-125 mg/dL
4. HbA1c between 5.7%~6.4%
5. Total Cholesterol≧160mg/dL or LDL-C≧100mg/dL Remark: Meet one of the (3)~(5) conditions is acceptable

Exclusion Criteria:

1. Pregnant and lactating women
2. Poor medication compliance
3. Abnormal liver function patients (ALT and AST value> 2 folds of normal value upper limit )
4. Abnormal renal function patients (creatinine value>1.5 mg/dL)
5. Abnormal gastrointestinal function patients (eg. gastrostomy, enterostomy, and diarrhea)
6. Sever comorbidity in the last 6 months. (eg. Brain stroke, myocardial infarction, and major trauma and surgery)
7. Using influence blood sugar, blood pressure, and blood lipid drugs (eg sex hormones, corticosteroids, H2 blockers, diuretics and Statin )
8. Diabetes patients
9. Other sever diseases ( malignant tumor and alzheimer's disease)
10. With inflammatory diseases, infectious disease, and severe immune deficiency ( eg. tuberculosis, AIDS, active pneumonia, systemic lupus erythematosus and rheumatoid arthritis)
11. Other influence blood sugar endocrine disease (eg. Hyperthyroidism, Acromegaly, Cushing's syndrome and Pheochromocytoma)

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of the change in lipid profile relative to baseline | 3 months
  Assessment of the change in Total Cholesterol(mg/dL), Triglyceride(mg/dL), low density lipoprotein (mg/dL) relative to baseline
Assessment of the change in lipid profile relative to baseline | 6 months
  Assessment of the change in Total Cholesterol(mg/dL), Triglyceride(mg/dL), low density lipoprotein (mg/dL) relative to baseline
Assessment of the change in inflammation index relative to baseline | 3 months
  Assessment of the change in TNF-alpha (pg/ml) and hs-CRP(pg/ml) relative to baseline
Assessment of the change in inflammation index relative to baseline | 6 months
  Assessment of the change in TNF-alpha (pg/ml) and hs-CRP(pg/ml) relative to baseline
Assessment of the change in HbA1C (%) relative to baseline | 3 months
  Assessment of the change in HbA1C (%) relative to baseline
Assessment of the change in HbA1C (%) relative to baseline | 6 months
  Assessment of the change in HbA1C (%) relative to baseline
Assessment of the change in fasting glucose (mg/dl) relative to baseline | 3 months
  Assessment of the change in fasting glucose (mg/dl) relative to baseline
Assessment of the change in fasting glucose (mg/dl) relative to baseline | 6 months
  Assessment of the change in fasting glucose (mg/dl) relative to baseline
Assessment of the change in liver function relative to baseline | 3 months
  Assessment of the change in ALT (U/L) and AST(U/L) relative to baseline
Assessment of the change in liver function relative to baseline | 6 months
  Assessment of the change in ALT (U/L) and AST(U/L) relative to baseline
Assessment of the change in renal function relative to baseline | 3 months
  Assessment of the change in Bun(mg/dL),Uric acid(mg/dL) and Creatinine(mg/dL) relative to baseline
Assessment of the change in renal function relative to baseline | 6 months
  Assessment of the change in Bun(mg/dL), Uric acid(mg/dL) and Creatinine(mg/dL) relative to baseline
Assessment of the change in Albumin (g/L) relative to baseline | 3 months
  Assessment of the change in Albumin (g/L) relative to baseline
Assessment of the change in Albumin (g/L) relative to baseline | 6 months
  Assessment of the change in Albumin (g/L) relative to baseline

CONTACTS AND LOCATIONS:
Overall Officials: TSE-HUNG HUANG, MD PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (2):
- Taiwan (2):
  - Center for traditional chinese medicine, Chang Gung Memorial Hospital, Gueishan Township, Taoyuan County
  - TSE-HUNG HUANG MD PhD, Keelung

IPD SHARING:
Plan to Share IPD: Undecided